CLINICAL TRIAL: NCT06594276
Title: Effectiveness of Local Instillation of Antibiotics Compared to Systemic Antibiotics, as Adjunct to Ultrasound Guided Aspiration in the Management of Breast Abscess; a Randomized Controlled Trial
Brief Title: Comparison of Efficacy in Treating Breast Abscess, With Systemic Antibiotics Against Local Instillation of Antibiotics Along With Ultrasound Guided Aspiration.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gujranwala medical college District Headquarters Hospital, Gujranwala (Other)
Responsible Party: Principal Investigator, Dr. Arslan Anwar, Post-Graduate Resident, Master of Surgery, General Surgery., Gujranwala medical college District Headquarters Hospital, Gujranwala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 341/GMC -23
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Abscess
Keywords: treatment of breast abscess

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle aspiration with systemic antibiotics (No Intervention)
- Needle aspiration with local instillation of antibiotics (Active Comparator)
  Interventions: Other: Local instillation of antibiotics

INTERVENTIONS:
Other: Local instillation of antibiotics — Systemic antibiotics are usually used with needle aspiration of breast abscess. However local instillation of antibiotics will be an in intervention in this study.
  Arms: Needle aspiration with local instillation of antibiotics

SUMMARY:
Breast abscess, marked by localized collection of pus, frequently follows mastitis. Its prevalence soars up to 16% in the developing world. It usually presents in lactating mothers but also develops in prepubertal females as well. Conventionally it has been treated by surgical incision and drainage with antibiotic coverage, whether oral, intramuscular or intravenous. This approach requires hospital stay and general anesthesia but also have complications like scarring and disfigurement. With the financial and emotional impacts of this technique , surgeons have opted needle aspiration of breast abscess as a standardized treatment. It has been very successful in the management of breast abscess as it spares the patients from long hospital stays and the cosmetic complications. It may require to repeat the procedure till the complete resolution of symptoms which can be effectively assessed by the clinical symptoms of the patient like redness of the skin, pain, tenderness and ultrasonographical evidence of pus accumulation. Systemic antibiotics are still frequently administered for prophylactic and therapeutic purposes. It has been shown in previous studies that systemic antibiotics may not be as effective as deemed earlier due to local pathogenesis. The use of local antibiotics is not a novel concept but a firmly established fact , whether its the earliest sterilization of the operative field or treating open wounds and fractures . Studies have shown great effect of local use of antibiotics in different scenarios and this may help in limit the use of antibiotics and providing the systemic bypass with maximum local impact. In patients of breast abscess, along with ultrasound guided aspiration the inclusion of locally injecting the antibiotics may reduce the frequency of procedure till the absolute resolution of symptoms and also markedly decrease the failure rate of this technique , which usually resorts to the conventional incision and drainage.

DETAILED DESCRIPTION:
A breast abscess is often characterized as a consequence of delayed or insufficient treatment following mastitis. The global prevalence of primary breast abscess in lactating women is estimated to be around 11%. In developing countries, where the quality of life and access to medical care may be limited, the prevalence of breast abscess tends to be higher. For instance, in Pakistan, the occurrence of breast abscess reaches up to 16%.

This condition typically arises due to local inflammation and/or infection of the terminal lactiferous ducts. Mastitis, a precursor to breast abscess, can be attributed to factors such as poor hygiene, inadequate breastfeeding practices, milk stasis, cracked nipples, and the colonization of Staphylococcus aureus. Patients with breast abscess typically present with a painful, tender, and either focally or diffusely swollen breast. It is noteworthy that breast abscesses can be broadly classified into lactational and non-lactational types, each contributing significantly to morbidity in adult women.

Several risk factors contribute to the development of both primary and recurrent lactational breast abscesses. These include increasing maternal age, obesity, primiparity, diabetes, smoking, and a history of mastitis. Additionally, rare predisposing factors encompass breast trauma, duct ectasia, fat necrosis, nipple piercing, and breast cancer.

Staphylococcus aureus remains the most common causative organism, although E. Coli and H. Influenza have also been identified. Of particular concern is the rising prevalence of Methicillin-Resistant Staphylococcus Aureus (MRSA).The traditional approach to managing breast abscesses involves Incision & Drainage (I&D) accompanied by antibiotic therapy. However, this method is primarily reserved for complicated cases with skin changes such as ulceration, necrosis, or recurrent abscesses. In recent years, needle aspiration has emerged as the preferred treatment for uncomplicated cases. Clinical examination and radiological assessments using ultrasound or CT are crucial for establishing the diagnosis. Notably, the breast surgery community increasingly adopts needle aspiration as a minimally invasive technique for cases where the abscess size is less than 5cm on ultrasound, and symptoms have persisted for up to 5 days. Needle aspiration offers advantages such as avoiding hospital stays,eliminating the need for general anesthesia, and allowing continued breast feeding. It also reduces the risk of complications like milk fistulae. Factors such as multiple dressings for wound care, pain, dissatisfaction with cosmetic results, and delayed healing with I&D contribute to the growing acceptance of aspiration as a suitable alternative.

Effective antimicrobial therapy is integral to the treatment of breast abscesses. Post I&D, antibiotic coverage is mandated for preventing Surgical Site Infection (SSI). The success of aspiration, similarly, hinges on judicious antimicrobial treatment. In an era marked by antibiotic resistance, providing effective and targeted antimicrobial therapy becomes crucial.

Studies highlight the benefits of local instillation of antibiotics, demonstrating promising results in preventing SSIs and managing wounds and abscesses. Local instillation not only provides bypasses systemic administration but also reduces the need for postoperative systemic antibiotics. The concentration of antibiotics at the local site is higher when instilled locally, as evidenced by in vitro studies showing a 100% kill rate after only 60 seconds of exposure to the antibiotic irrigating solution. With advancement and diversity in the field of surgery, it is adapting to minimally invasive procedures with efficient out comes and conserving cosmetics. Aspiration for breast abscesses is replacing the conventional I&D to provide better care, fewer complications and better cosmetic results. In stemming the rise of resistance patterns antimicrobial stewardship has become surgical obligation. Some studies show that aspiration of the breast abscess with systemic antibiotics has a success rate of up to 94%, around 50%- 60% of the cases are recovered after single aspiration while some 20%-30% required a second time and rest needed multiple aspirations. The use of local instillation of antibiotics adjunct to aspiration in management of breast abscess may help limit the number of aspirations and recurrence, providing better cure and healing time for the patients. Abscess wall and edema makes it take longer to achieve MIC (minimal inhibitory concentration) than the local instillation. It can also help to limit the use of systemic antibiotics, and promote continued breast feeding. Combined they can not only cut down the morbidity but also prove to be better in treating the breast abscess and a key step against the emerging antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

- Female gender Age range 14-60 years Lactating or non-lactating Clinical signs : erythema, tenderness, fever, fluctuation

Exclusion Criteria:

Patients refusal Male gender Acute mastitis Malignant lesion (inflammatory carcinoma) Antibioma Draining abscess/Sinus Skin ulcers / gangrene Diagnosed case of Tuberclosis H.I.V

-

Ages: 14 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 104 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy | From enrollment to the end of treatment at 9 days
  The number of times the procedure is repeated till the resolution of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Gujranwala Medical College, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Barron AU, Luk S, Phelan HA, Williams BH. Do acute-care surgeons follow best practices for breast abscess management? A single-institution analysis of 325 consecutive cases. J Surg Res. 2017 Aug;216:169-171. doi: 10.1016/j.jss.2017.05.013. Epub 2017 May 10. PMID 28807202
- [Background] Afridi SP, Alam SN, Ainuddin S. Aspiration of breast abscess through wide bore 14-gauge intravenous cannula. J Coll Physicians Surg Pak. 2014 Oct;24(10):719-21. doi: 10.2014/JCPSP.719721. PMID 25327913